CLINICAL TRIAL: NCT05028582
Title: A Randomized tRial Employing topiCal roflumilasT Foam to Treat Scalp Psoriasis (ARRECTOR)
Brief Title: Topical Roflumilast to Treat Scalp and Body Psoriasis (ARRECTOR)
Acronym: ARRECTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-154-309
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Foam 0.3% (Active Comparator): Participants with plaque psoriasis of the scalp and body applied roflumilast foam 0.3% once daily (qd) for 8 weeks.
  Interventions: Drug: Roflumilast Foam 0.3%
- Vehicle Foam (Placebo Comparator): Participants with plaque psoriasis of the scalp and body applied vehicle foam qd for 8 weeks.
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Roflumilast Foam 0.3% — Roflumilast foam 0.3%
  Other Names: ARQ-154 0.3%
  Arms: Roflumilast Foam 0.3%
Drug: Vehicle Foam — Vehicle foam matched to roflumilast 0.3% foam.
  Arms: Vehicle Foam

SUMMARY:
This was a parallel group, double blind, vehicle-controlled study to assess the safety and efficacy of roflumilast (ARQ-154) 0.3% foam vs vehicle foam applied once daily (qd) for 8 weeks by participants with plaque psoriasis of the scalp and body.

ELIGIBILITY:
Inclusion Criteria:

* For adult subjects: Participants legally competent to read, write, and sign and give informed consent. For adolescent subjects: Informed consent of a parent(s) or legal guardian, and assent by the subjects, as required by local laws.
* Males and females ages 12 years and older (inclusive) at the time of consent or assent.
* Scalp psoriasis with a Scalp-Investigator Global Assessment of Disease (S IGA) severity of at least Moderate ('3') at Baseline.
* Extent of scalp psoriasis involving ≥ 10% of the total scalp at Baseline.
* A Psoriasis Scalp Severity Index (PSSI) of at least 6 at Baseline.
* An IGA of body (i.e., non-scalp) psoriasis (B-IGA) of at least Mild ('2') at Baseline.
* A PASI score of at least 2 (excluding palms and soles) at Baseline.
* Clinical diagnosis of psoriasis vulgaris of at least 6 months duration at Screening as determined by the Investigator. Stable disease for the past 4 weeks.
* Total overall psoriasis involvement on scalp and non-scalp areas ≤ 25% BSA (not including palms/soles) at Baseline. Total non-scalp BSA should not exceed 20%.
* Female subject of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and negative urine pregnancy test at Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception or a barrier method of contraception throughout the study according to Contraception Requirements for the protocol.
* Females of non-childbearing potential must either be premenarchal, post-menopausal with spontaneous amenorrhea for at least 12 months (post-menopausal status will be confirmed with FSH testing) or have undergone surgical sterilization according to Contraception Requirements for the protocol. Prepubescent females must agree to be abstinent during the study.
* Subjects in good health as judged by the Investigator, based on medical history, physical examination, vital signs, serum chemistry labs, hematology values, and urinalysis.

Exclusion Criteria:

* Subjects who cannot discontinue treatment with therapies for the treatment of psoriasis vulgaris prior to the Baseline visit and during the study.
* Planned excessive exposure to treated area(s) to either natural or artificial sunlight, tanning bed, or other LED.
* Previous treatment with ARQ-151 or ARQ-154.
* Females who are pregnant, wishing to become pregnant during the study, or are breast feeding.
* Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
* Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members residing in the same household of enrolled subjects.
* Any condition that in the Investigator's assessment would preclude the subject from participating in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (49):
- United States (36):
  - Arcutis Biotherapeutics Clinical Site 01, Scottsdale, Arizona
  - Arcutis Biotherapeutics Clinical Site 50, Beverly Hills, California
  - Arcutis Biotherapeutics Clinical Site 45, Encinitas, California
  - Arcutis Biotherapeutics Clinical Site 64, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 72, Santa Ana, California
  - Arcutis Biotherapeutics Clinical Site 21, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 33, Clearwater, Florida
  - Arcutis Biotherapeutics Clinical Site 42, Coral Gables, Florida
  - Arcutis Biotherapeutics Clinical Site 57, Delray Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 31, North Miami Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 05, Orlando, Florida
  - Arcutis Biotherapeutics Clinical Site 65, Sanford, Florida
  - Arcutis Biotherapeutics Clinical Site 12, Tampa, Florida
  - Arcutis Biotherapeutics Clinical Site 22, Plainfield, Illinois
  - Arcutis Biotherapeutics Clinical Site 10, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 15, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 04, Lake Charles, Louisiana
  - Arcutis Biotherapeutics Clinical Site 02, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 28, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 20, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 14, New Brighton, Minnesota
  - Arcutis Biotherapeutics Clinical Site 44, Saint Joseph, Missouri
  - Arcutis Biotherapeutics Clinical Site 34, East Windsor, New Jersey
  - Arcutis Biotherapeutics Clinical Site 51, Rochester, New York
  - Arcutis Biotherapeutics Clinical Site 63, The Bronx, New York
  - Arcutis Biotherapeutics Clinical Site 23, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 25, Portland, Oregon
  - Arcutis Biotherapeutics Clinical Site 27, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 06, Knoxville, Tennessee
  - Arcutis Biotherapeutics Clinical Site 13, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 11, Austin, Texas
  - Arcutis Biotherapeutics Clinical Site 41, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 54, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 24, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 07, West Jordan, Utah
  - Arcutis Biotherapeutics Clinical Site 17, Norfolk, Virginia
- Canada (13):
  - Arcutis Biotherapeutics Clinical Site 35, Calgary, Alberta
  - Arcutis Biotherapeutics Clinical Site 37, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 47, Winnepeg, Manitoba
  - Arcutis Biotherapeutics Clinical Site 43, Fredericton, New Brunswick
  - Arcutis Biotherapeutics Clinical Site 38, Ajax, Ontario
  - Arcutis Biotherapeutics Clinical Site 16, London, Ontario
  - Arcutis Biotherapeutics Clinical Site 29, Mississauga, Ontario
  - Arcutis Biotherapeutics Clinical Site 30, North Bay, Ontario
  - Arcutis Biotherapeutics Clinical Site 32, Peterborough, Ontario
  - Arcutis Biotherapeutics Clinical Site 71, Toronto, Ontario
  - Arcutis Biotherapeutics Clinical Site 36, Waterloo, Ontario
  - Arcutis Biotherapeutics Clinical Site 49, Windsor, Ontario
  - Arcutis Biotherapeutics Clinical Site 09, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gooderham MJ, Alonso-Llamazares J, Bagel J, Bhatia N, Bukhalo M, DuBois J, Ferris LK, Green L, Kircik LH, Lockshin B, Loo WJ, Papp KA, Soung J, Seal MS, Snyder S, Kato S, Krupa D, Burnett P, Berk DR, Chu DH. Roflumilast Foam, 0.3%, for Psoriasis of the Scalp and Body: The ARRECTOR Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2025 Jul 1;161(7):698-706. doi: 10.1001/jamadermatol.2025.1136. PMID 40332898

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 53 study centers in the US and Canada.
Groups:
- Roflumilast Foam 0.3%: Participants with plaque psoriasis of the scalp and body applied roflumilast foam 0.3% qd for 8 weeks.
Period: Overall Study
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Started | 281 | 151
Completed | 250 | 126
Not Completed | 31 | 25
Not completed — Lost to Follow-up | 11 | 9
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Adverse Event | 5 | 2
Not completed — Miscellaneous | 3 | 2
Not completed — Lack of Efficacy | 3 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam | Total
Number analyzed (Participants) | 281 | 151 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.93) | 45.0 (14.33) | 47.3 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 91 | 243
  Male | 129 | 60 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 28 | 76
  Not Hispanic or Latino | 224 | 121 | 345
  Unknown or Not Reported | 9 | 2 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American-Indian or Alaska Native | 0 | 3 | 3
  Asian | 26 | 4 | 30
  Black or African-American | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  White | 225 | 129 | 354
  Other | 11 | 7 | 18
  More than One Race | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Scalp Investigator Global Assessment (S-IGA) "Success" at Week 8
Description: The percentage of participants with S-IGA success at Week 8 is presented. Success is defined as an IGA score of 'clear' or 'almost clear' plus a 2-point improvement from baseline at Week 8. This global assessment scale has five severity grades reported from 0-4 and defined as Clear (0), Almost Clear (1), Mild (2), Moderate (3), Severe (4), with higher scores indicative of greater symptom severity.
Time Frame: Week 8
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 66.4 [59.62 to 72.56] | 27.8 [20.12 to 37.10]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; S-IGA Success at Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio, log = 5.19, 97.5% CI 2-sided [2.90 to 9.31] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

2. Primary Outcome: Achievement of Body Investigator Global Assessment (B-IGA) Success at Week 8
Description: The percentage of participants with B-IGA success at Week 8 is presented. Success is defined as an IGA score of 'clear' or 'almost clear' plus a 2-point improvement from baseline at Week 8. This global assessment scale has five severity grades reported from 0-4 and defined as Clear (0), Almost Clear (1), Mild (2),Moderate (3), Severe (4), with higher scores indicative of greater symptom severity.
Time Frame: Week 8
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 45.5 [38.87 to 52.33] | 20.1 [13.55 to 28.81]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; B-IGA Success at Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 3.17, 97.5% CI 2-sided [1.75 to 5.73] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

3. Secondary Outcome: Achievement of Scalp Itch-Numeric Rating Score (SI-NRS ) Success at Week 2
Description: The percentage of participants with SI-NRS success at Week 2 is presented. Success is defined as a ≥ 4-point improvement from baseline weekly in weekly average SI-NRS in participants with weekly average baseline SI-NRS score ≥4. SI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale ranges from 0 ("no itch") to 10 ("worst imaginable itch"), with higher scores indicative of greater symptom severity.
Time Frame: Week 2
Population: All randomized participants with weekly average baseline SI-NRS ≥4 are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 203 | 123
percentage of participants | 25.2 [18.96 to 32.63] | 8.0 [3.90 to 15.55]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Other — SI-NRS Success at Week 4; p = 0.0005, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.67, 97.5% CI 2-sided [1.60 to 13.62] — Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data

4. Secondary Outcome: Achievement of SI-NRS Success at Week 4
Description: The percentage of participants with SI-NRS success at Week 4 is presented. Success is defined as a ≥ 4-point improvement from baseline weekly in weekly average SI-NRS in participants with weekly average baseline SI-NRS score ≥4. SI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale ranges from 0 ("no itch") to 10 ("worst imaginable itch"), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants with weekly average baseline SI-NRS ≥4 are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 203 | 123
percentage of participants | 46.2 [38.32 to 54.22] | 16.8 [10.40 to 26.04]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; SI-NRS Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.39, 97.5% CI 2-sided [2.01 to 9.55] — Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data

5. Secondary Outcome: Achievement of SI-NRS Success at Week 8
Description: The percentage of participants with SI-NRS success at Week 8 is presented. Success is defined as a ≥ 4-point improvement from baseline weekly in weekly average SI-NRS in participants with weekly average baseline SI-NRS score ≥4. SI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale ranges from 0 ("no itch") to 10 ("worst imaginable itch"), with higher scores indicative of greater symptom severity.
Time Frame: Week 8
Population: All randomized participants with weekly average baseline SI-NRS ≥4 are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 203 | 123
percentage of participants | 65.3 [57.26 to 72.58] | 30.3 [21.38 to 40.91]
Statistical Analysis 1: Comparison: Vehicle Foam; Test type: Other — SI-NRS Success at Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 5.41, 97.5% CI 2-sided [2.49 to 11.78] — Stratified by pooled study site, baseline S IGA, and baseline B-IGA with multiple imputation to handle missing data

6. Secondary Outcome: Change From Baseline in SI-NRS Score at Day 1
Description: SI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale ranges from 0 ("no itch") to 10 ("worst imaginable itch"), with higher scores indicative of greater symptom severity. A negative change from baseline indicates symptom improvement, and vice versa.
Time Frame: Day 1
Population: All randomized participants with average, weekly SI-NRS ≥4 at baseline are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
score on a scale | -0.44 (0.120) | -0.09 (0.149)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — SI-NRS Change from Baseline Day 1; p = 0.0164, ANCOVA; ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score; LS Mean Difference = -0.35, 97.5% CI 2-sided [-0.68 to -0.02] — ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score

7. Secondary Outcome: Change From Baseline in SI-NRS Score at Day 3
Description: as for outcome 6
Time Frame: Day 3
Population: All randomized participants are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
score on a scale | -1.11 (0.133) | -0.36 (0.165)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — SI-NRS Change from Baseline Day 1; p < 0.0001, ANCOVA; ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score; LS Mean Difference = -0.76, 97.5% CI 2-sided [-1.12 to -0.39] — ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score

8. Secondary Outcome: Change From Baseline in SI-NRS Score at Week 1
Description: as for outcome 6
Time Frame: Week 1
Population: All randomized participants are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
score on a scale | -1.08 (0.121) | -0.53 (0.151)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — Change from Baseline in Weekly SI-NRS at Week 1; p = 0.0002, ANCOVA; ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score; LS Mean Difference = -0.55, 97.5% CI 2-sided [-0.87 to -0.22] — ANCOVA terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline SI-NRS score

9. Secondary Outcome: Achievement of WI-NRS (Worst Itch-Numeric Rating Score) Success at Week 8
Description: WI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale is from 0 ("no itch") to 10 ("worst imaginable itch"). Success is defined as achievement of a ≥ 4-point improvement from baseline in participants with a baseline WI-NRS pruritus score of ≥ 4.
Time Frame: Week 8
Population: All randomized participants with average, weekly WI-NRS ≥4 at baseline are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 203 | 110
percentage of participants | 63.1 [54.97 to 70.59] | 30.1 [20.69 to 41.44]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3%; Test type: Other — WI-NRS Success at Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA; Odds Ratio (OR) = 4.14, 97.5% CI 2-sided [2.01 to 8.52] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA

10. Secondary Outcome: Achievement of a 75% Reduction From Baseline in Psoriasis Area and Severity Index (PASI-75)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. A decrease from baseline indicates symptom improvement, and vice versa.
Time Frame: Week 8
Population: All randomized participants are included, with multitple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 50.1 [43.24 to 56.91] | 16.8 [10.77 to 25.15]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3%; Test type: Superiority — PASI-75 at Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 5.42, 97.5% CI 2-sided [2.73 to 10.75] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

11. Secondary Outcome: Change From Baseline in Psoriasis Symptoms Diary (PSD) Aggregate Score of Itching, Pain, and Scaling (Questions 1, 9, and 11)
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. The aggregate Itching, Pain, and Scaling score ranges from 0 to 30; the change from baseline in aggregate score was assessed per protocol only in adult participants.
Time Frame: Week 8
Population: All randomized participants ≥18 years of age are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 274 | 148
score on a scale | -10.87 (0.546) | -5.75 (0.698)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — PSD Aggregate Score Change at Week 8; p < 0.0001, ANCOVA; Covariate terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA and baseline PSD aggregate score & multiple imputation of missing data; LS Mean Difference = -5.12, 97.5% CI 2-sided [-6.64 to -3.60] — Covariate terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA and baseline PSD aggregate score & multiple imputation of missing data

12. Secondary Outcome: Percentage of Participants Achieving PSD Itching (Question 1) Score of 0 at Week 8
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. The Scaling score ranges from 0 to 10.
Time Frame: Week 8
Population: All randomized participants ≥18 years of age are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 274 | 148
percentage of participants | 31.7 [25.63 to 38.58] | 10.0 [5.55 to 17.32]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3%; Test type: Superiority — PSD Itching Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.59, 97.5% CI 2-sided [2.10 to 10.04] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

13. Secondary Outcome: Percentage of Participants Achieving PSD Pain (Question 9) Score of 0 at Week 8
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. The Pain score ranges from 0 to 10.
Time Frame: Week 8
Population: All randomized participants ≥18 years of age are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 274 | 148
percentage of participants | 64.9 [58.03 to 71.24] | 40.3 [31.36 to 49.95]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — PSD Pain Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 3.23, 97.5% CI 2-sided [1.83 to 5.68] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

14. Secondary Outcome: Percentage of Participants Achieving PSD Scaling (Question 11) Score of 0 at Week 8
Description: as for outcome 12
Time Frame: Week 8
Population: All randomized participants ≥18 years of age are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 274 | 148
percentage of participants | 41.5 [34.86 to 48.54] | 13.6 [8.26 to 21.59]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — PSD Scaling Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.56, 97.5% CI 2-sided [2.28 to 9.08] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

15. Secondary Outcome: Percentage of Participants Achieving PSD Total Score of 0 at Week 8
Time Frame: Week 8
Population: All randomized participants ≥18 years of age are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 274 | 148
percentage of participants | 19.6 [14.65 to 25.82] | 7.1 [3.50 to 13.79]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Other — PSD Total Score 0 at Week 8; p = 0.0012, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA; Odds Ratio (OR) = 3.27, 97.5% CI 2-sided [1.39 to 7.68] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA

16. Secondary Outcome: Achievement of a 75% Reduction From Baseline in Psoriasis Scalp Severity Index (PSSI) Score (PSSI-75)
Description: The PSSI combines the assessment of the severity of scalp lesions and the area of scalp affected into a single score in the range 0 (no disease) to 72 (maximal disease). PSSI combines the assessment of the severity of scalp lesions and the area of scalp affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Time Frame: Week 8
Population: All randomized participants are included, with multiple imputation of missing data..
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 70.9 [64.27 to 76.70] | 31.3 [23.15 to 40.72]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — PSSI-75 at Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S IGA, and baseline B IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 5.40, 97.5% CI 2-sided [2.98 to 9.77] — Stratified by pooled study site, baseline S IGA, and baseline B IGA with multiple imputation to handle missing data

17. Secondary Outcome: Achievement of S-IGA Score of 'Clear' at Week 8
Description: The percentage of participants with S-IGA score of 0 Week 8 is presented. This global assessment scale has five severity grades reported from 0-4 and defined as Clear (0), Almost Clear (1), Mild (2), Moderate (3), Severe (4), with higher scores indicative of greater symptom severity.
Time Frame: Week 8
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 40.0 [33.47 to 46.81] | 9.1 [4.88 to 16.18]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — S-IGA Clear at Week 8; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 6.77, 97.5% CI 2-sided [3.04 to 15.05] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

18. Secondary Outcome: Achievement of S-IGA Success at Week 2
Description: The percentage of participants with S-IGA success at Week 2 is presented. Success is defined as an IGA score of 'clear' or 'almost clear' plus a 2-point improvement from baseline. This global assessment scale has five severity grades reported from 0-4 and defined as Clear (0), Almost Clear (1), Mild (2), Moderate (3), Severe (4), with higher scores indicative of greater symptom severity.
Time Frame: Week 2
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 30.4 [24.62 to 36.92] | 11.7 [6.90 to 19.20]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — S-IGA Success Week 2; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.10, 97.5% CI 2-sided [1.84 to 9.13] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

19. Secondary Outcome: Achievement of S-IGA Success at Week 4
Description: The percentage of participants with S-IGA success at Week 4 is presented. Success is defined as an IGA score of 'clear' or 'almost clear' plus a 2-point improvement from baseline. This global assessment scale has five severity grades reported from 0-4 and defined as Clear (0), Almost Clear (1), Mild (2), Moderate (3), Severe (4), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
percentage of participants | 53.8 [47.00 to 60.46] | 19.5 [13.09 to 27.95]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — S-IGA Success at Week 4; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data; Odds Ratio (OR) = 4.82, 97.5% CI 2-sided [2.62 to 8.84] — Stratified by pooled study site, baseline S-IGA, and baseline B-IGA with multiple imputation to handle missing data

20. Secondary Outcome: Change From Baseline in PASI Score at Week 2
Description: as for outcome 10
Time Frame: Week 2
Population: All randomized participants are included, with multiple imputation of missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 281 | 151
score on a scale | -2.31 (0.157) | -1.03 (0.193)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Test type: Superiority — Change from Baseline in PASI Week 2; p < 0.0001, ANCOVA; Covariate terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline PASI score & multiple imputation to handle missing data; LS Mean Difference = -1.28, 97.5% CI 2-sided [-1.71 to -0.85] — Covariate terms of treatment, pooled study site, baseline S-IGA, baseline B-IGA, and baseline PASI score & multiple imputation to handle missing data

ADVERSE EVENTS:
Time Frame: Up to ~12 weeks (8 weeks of treatment + 4 weeks of follow-up)
Description: All treated participants are included.
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/151
Serious Adverse Events (participants affected / at risk) | 2/281 | 1/151
Other Adverse Events (participants affected / at risk) | 0/281 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Foam 0.3% (N=281) | Vehicle Foam (N=151)
Bipolar disorder (Psychiatric disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT05028582/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05028582/SAP_001.pdf